CLINICAL TRIAL: NCT01836692
Title: Isotoxic Intensity Modulated Radiotherapy (IMRT) in Stage III Non Small Cell Lung Cancer (NSCLC) - A Feasibility Study
Acronym: Isotoxic-IMRT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Prof Corinne Faivre-Finn (Other)
Collaborators: Cancer Research UK (Other); British Lung Foundation (Other); Sheffield Teaching Hospitals NHS Foundation Trust (Other); Belfast Health and Social Care Trust (Other); The Leeds Teaching Hospitals NHS Trust (Other); Cambridge University Hospitals NHS Foundation Trust (Other); Royal Marsden NHS Foundation Trust (Other); East and North Hertfordshire NHS Trust (Other Government)
Responsible Party: Sponsor-Investigator, Prof Corinne Faivre-Finn, Prof Corinne Faivre-Finn, Consultant Clinical Oncologist, The Christie NHS Foundation Trust
Organization: The Christie NHS Foundation Trust (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 11_DOG07_136
Record Dates: First submitted 2013-04-12; First posted 2013-04-22 (Estimated); Last update posted 2018-10-31 (Actual); Status verified 2018-10

CONDITIONS: Non Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Thoracic radiotherapy (Experimental): Intensity Modulated Radiotherapy treatment (delivered twice daily on consecutive weekdays over 4.5 weeks)
  Interventions: Radiation: Intensity Modulated Radiotherapy treatment

INTERVENTIONS:
Radiation: Intensity Modulated Radiotherapy treatment — Intensity Modulated Radiotherapy treatment

SUMMARY:
This study is for patients having a course of chest radiotherapy treatment after receiving chemotherapy for the treatment of non-small cell lung cancer. Patients with non-small cell lung cancer have a risk of the tumour in the lung recurring or progressing after treatment.

In this study, we will investigate:

* whether giving a more targeted and individualised type of chest irradiation or radiotherapy to the lung tumour (known as Isotoxic IMRT), is practical and whether it causes side effects which can be tolerated
* whether this new method of delivering the radiotherapy can reduce the risk of the tumour in the lung recurring or progressing
* whether survival can be improved by using this new radiotherapy method

The dose of chest irradiation will be calculated specifically to suit patient's body shape, the position of the lung cancer, and how close healthy tissues are to the tumour. Radiotherapy will be delivered twice a day over a maximum period of 4.5 weeks. The duration of treatment will vary individually according to the delivered dose to the tumour area.

DETAILED DESCRIPTION:
Background:

Approximately 12,000 patients are diagnosed with stage III NSCLC in the UK each year and their survival is ~15% at 5 years. As the majority of patients are not suitable for the gold standard treatment (concurrent chemo-radiotherapy (CTRT), novel strategies integrating radiotherapy (RT) technological advances and radiobiological knowledge need to be evaluated in patients treated with the alternative treatment option, sequential CTRT. There is solid evidence that improving local control in lung cancer leads to increased survival. Strategies to improve local control in stage III NSCLC include dose escalation and individualisation which are limited by the dose delivered to surrounding normal tissues. We hypothesise that this will be facilitated by the use of IMRT.

Objectives:

To demonstrate the feasibility of delivering isotoxic RT using IMRT and hyperfractionated accelerated RT in stage III NSCLC patients who are not suitable for concurrent CTRT.

Endpoints:

Primary endpoint: Delivery of isotoxic IMRT to dose >60 Gy EQD2 (total biologically equivalent in 2 Gy fraction).

Secondary endpoints: Estimation of the suitability for lung isotoxic IMRT, estimation of proportion of patients with acute grade 3+ non haematological toxicity, estimation of late toxicity, estimation of local control/overall survival and development of a robust Quality Assurance (QA) process for lung IMRT.

Design:

Prospective multicentre, non-randomised feasibility study with early stopping rules.

35 patients will be recruited in this prospective multicentre feasibility study. Stopping rules are in place to ensure the safety of patients. We estimate that this regimen would be of added value to a national randomised phase II trial if 80% of the patients can be planned to a dose >60 Gy EQD2.

Intervention:

Patients with stage III NSCLC, PS 0-2, not suitable for concurrent CTRT, will be treated with individualised doses of radiation based on pre-specified normal tissue doses (spinal cord, brachial plexus, lung tissue, heart and great vessels/proximal bronchial tree). Radiotherapy will be delivered twice-daily over a maximum period of 4.5 weeks using IMRT and the dose of radiation will be increased until one or more of the organs at risk tolerance or the maximum dose of 79.2 Gy is reached.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed NSCLC
* Inoperable Stage III disease (T3N1-3, any T4, any N2 -3) confirmed by PET scanning, mediastinoscopy or thoracoscopy
* Patients treated with at least 2 cycles of platinum based induction chemotherapy and able to start radiotherapy within 5 weeks of the last cycle of chemotherapy
* Tumour judged inoperable by a lung MDT
* Age 18+, no upper age limit
* Performance status (PS) - ECOG 0-2. Patients with PS 2 whose general condition is explained by disease can be included at the discretion of the local investigator. Patients with PS 2 as a result of co-morbid conditions will be excluded
* Patient considered suitable for radical RT
* Tumour that can be encompassed within a radical RT treatment volume (MLD expected to be <20Gy)

Exclusion Criteria:

* Patients suitable for standard concurrent CTRT
* Patients only suitable for radical RT due to PS and co-morbidities

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2014-04 (Actual); Primary Completion 2016-10 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
The number of participants treated with isotoxic RT (to dose >60 Gy EQD2) using IMRT & hyperfractionated accelerated RT. | Stage 1 (12 months) - after 19 patients have been treated with isotoxic IMRT
  Radiotherapy treatment plans & OAR tolerance doses will be analysed to assess the feasibility of delivering the proposed treatment.

SECONDARY OUTCOMES:
The number of participants from the study population who are suitable to receive isotoxic IMRT treatment. | 12 months
  Stage 1 - if 13/19 patients can be planned to a dose of >60 Gy EQD2 the study will proceed to stage 2 and recruit a further 16 patients. Assessed via RT planning data.
The number of participants treated with isotoxic IMRT who experience grade 3+ pulmonary toxicity | 12 months
  Stage 1 - if <3/19 participants experience grade 3+ acute pulmonary toxicity the study will proceed to stage 2 and recruit a further 16 patients. Assessed via toxicity data.
The number of participants treated with isotoxic IMRT who experience acute grade 3+ non haematological toxicity & other late toxicities | 12 months
  To assess via toxicity data, the number of patients who experience grade 3+ non haematological toxicities and other late toxicities
Number of participants whose disease is controlled locally & overall survival rates | Follow up visits every 4 months for 2 years & then 6 monthly for up to 5 years
  After completion of radiotherapy treatment regular follow up will continue and data on long term toxicity, local control and survival will be collected.

CONTACTS AND LOCATIONS:
Overall Officials: Corinne Faivre-Finn, MD PhD, Principal Investigator — The Christie NHS Foundation Trust
Locations (7):
- United Kingdom (7):
  - Belfast Health & Social Care NHS Trust - Northern Ireland Cancer Centre, Belfast
  - Cambridge University Hospitals NHS Foundation Trust - Addenbrookes Hospital, Cambridge
  - Beatson West of Scotland Cancer Centre, Glasgow
  - Leeds Teaching Hospitals NHS Trust - St James's University Hospital, Leeds
  - The Christie NHS Foundation Trust, Manchester
  - Sheffield Teaching Hospitals NHS Foundation Trust - Weston Park Hospital, Sheffield
  - The Royal Marsden NHS Foundation Trust, Surrey

REFERENCES:
- [Derived] Haslett K, Franks K, Hanna GG, Harden S, Hatton M, Harrow S, McDonald F, Ashcroft L, Falk S, Groom N, Harris C, McCloskey P, Whitehurst P, Bayman N, Faivre-Finn C. Protocol for the isotoxic intensity modulated radiotherapy (IMRT) in stage III non-small cell lung cancer (NSCLC): a feasibility study. BMJ Open. 2016 Apr 15;6(4):e010457. doi: 10.1136/bmjopen-2015-010457. PMID 27084277